CLINICAL TRIAL: NCT04496427
Title: A Single-center, Long-term, Observational Study to Determine the Efficacy and Safety of Potenfill for Temporary Penile Enhancement
Brief Title: Observational Study to Determine the Efficacy and Safety of Potenfill for Temporary Penile Enhancement
Status: Completed | Type: Observational
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Other Study IDs: MT05-KR19PGE1101
Record Dates: First submitted 2020-07-27; First posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Penile Enhancement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study to determine the efficacy and safety of Potenfill for temporary penile enhancement.

The pivotal study of Potenfill has already been completed and this observational study determines the long-term efficacy and safety for up to 24 months in subjects who have been participated and treated in the pivotal study.

ELIGIBILITY:
Inclusion Criteria:

* Males over 19 and under 65 who have participated in the previous clinical investigation (pivotal) and were treated with the investigational medical device and completed all the anticipated visits.

Exclusion Criteria:

* Subjects who have received any procedures or surgeries (penile enhancement procedure, HA filler, collagen, etc.) in the penile area from the time after the participation of the previous clinical investigation (pivotal) and before the screening for this clinical investigation.
* Subjects deemed as ineligible to participate by the investigator

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males over 19 and under 65 who have participated in the previous clinical investigation (pivotal) and were treated with the investigational medical device and completed all the anticipated visits.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the appearance of penis assessed by the Subject Satisfaction at 18 months after treatment with Potenfill compared to baseline | 18 months
  Satisfaction with the physical appearance of the penis as assessed by the subject at 18 months after application of the investigational medical device compared to baseline. The Subject Satisfaction score ranges from 1 (extremely unsatisfied) to 7 (extremely satisfied).
Satisfaction with the appearance of penis assessed by the Subject Satisfaction at 24 months after treatment with Potenfill compared to baseline | 24 months
  Satisfaction with the physical appearance of the penis as assessed by the subject at 24 months after application of the investigational medical device compared to baseline. The Subject Satisfaction score ranges from 1 (extremely unsatisfied) to 7 (extremely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Kangdong Sacred Heart Hospital, Seoul, Gangdong-gu, South Korea